CLINICAL TRIAL: NCT03449667
Title: Cryoanalgesia to Treat Post-Amputation Phantom Limb Pain: A Multicenter, Randomized, Double-Masked, Placebo-Controlled, Definitive Human Subjects Clinical Trial
Brief Title: Cryoanalgesia to Treat Post-Amputation Phantom Limb Pain: A Department of Defense Funded Multicenter Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Brian M. Ilfeld, MD, MS, Professor of Anesthesiology, In Residence, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CRYO for Phantom Pain (DoD); W81XWH-17-2-0051 (Other Grant/Funding Number: Peer Reviewed Medical Research Program (PRMRP)); PR160263 (Other Grant/Funding Number: Department of Defense Congressionally Directed Medical Research Programs)
Record Dates: First submitted 2018-02-22; First posted 2018-02-28 (Actual); Results first posted 2023-02-17 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Post-Amputation Phantom Limb Pain

STUDY DESIGN:
Intervention Model Description: The primary endpoint at 4 months following the initial treatment will utilize a parallel group study design; however, an optional crossover is offered to subjects following this time point.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: All individuals will be masked to treatment with the exception of the anesthesiologist administering the procedure who will choose which probe to use: the functional or sham. Of note, this individual could not be masked to treatment since the cryoneurolysis ice ball is visualized on ultrasound; and, the practitioner would see a lack of ice ball formation for the sham probes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Cryoneurolysis first, then optional sham crossover treatment (Active Comparator): Initial treatment: Cryoneurolysis of the femoral and sciatic nerves (or their distal counterparts) in the residual limb: The cryoneurolysis device will be triggered using 3 cycles of 2-minute gas activation separated by 1-minute defrost periods. For active probes, the nitrous oxide will be deployed to the tip where a drop in temperature to -70°C will result in cryoneurolysis.
  Optional sham crossover treatment: Sham cryoneurolysis of the femoral and sciatic nerves (or their distal counterparts) in the residual limb: The cryoneurolysis device will be triggered using 3 cycles of 2-minute gas activation separated by 1-minute defrost periods. However, for sham probes, the nitrous oxide is not deployed to the tip and therefore there is no drop in temperature resulting in cryoneurolysis.
  Interventions: Device: Cryoneurolysis; Device: Sham Comparator
- Sham Comparator first, then optional cryoneurolysis treatment (Sham Comparator): Initial treatment: Sham cryoneurolysis of the femoral and sciatic nerves (or their distal counterparts) in the residual limb: The cryoneurolysis device will be triggered using 3 cycles of 2-minute gas activation separated by 1-minute defrost periods. However, for sham probes, the nitrous oxide is not deployed to the tip and therefore there is no drop in temperature resulting in cryoneurolysis.
  Optional cryoneurolysis treatment: Cryoneurolysis of the femoral and sciatic nerves (or their distal counterparts) in the residual limb: The cryoneurolysis device will be triggered using 3 cycles of 2-minute gas activation separated by 1-minute defrost periods. For active probes, the nitrous oxide will be deployed to the tip where a drop in temperature to -70°C will result in cryoneurolysis.
  Interventions: Device: Cryoneurolysis; Device: Sham Comparator

INTERVENTIONS:
Device: Cryoneurolysis — Cryoneurolysis of the femoral and sciatic nerves (or their distal counterparts) in the residual limb: The cryoneurolysis device will be triggered using 3 cycles of 2-minute gas activation separated by 1-minute defrost periods. For active probes, the nitrous oxide will be deployed to the tip where a drop in temperature to -70°C will result in cryoneurolysis.
  Other Names: Cryoanalgesia
Device: Sham Comparator — Sham cryoneurolysis of the femoral and sciatic nerves (or their distal counterparts) in the residual limb: The cryoneurolysis device will be triggered using 3 cycles of 2-minute gas activation separated by 1-minute defrost periods. However, for sham probes, the nitrous oxide is not deployed to the tip and therefore there is no drop in temperature resulting in cryoneurolysis.
  Other Names: placebo, control

SUMMARY:
When a limb is severed, pain perceived in the part of the body that no longer exists often develops and is called "phantom limb" pain. Unfortunately, phantom pain goes away in only 16% of afflicted individuals, and there is currently no reliable definitive treatment. The exact reason that phantom limb pain occurs is unclear, but when a nerve is cut-as happens with an amputation-changes occur in the brain and spinal cord that actually increase with worsening phantom pain. These abnormal changes may often be corrected by putting local anesthetic-called a "nerve block"-on the injured nerve, effectively keeping any "bad signals" from reaching the brain with a simultaneous resolution of the phantom limb pain. However, when the nerve block resolves after a few hours, the phantom pain returns. But, this demonstrates that the brain abnormalities-and phantom pain-that occur with an amputation are not necessarily fixed, and may be dependent upon the "bad" signals being sent from the injured nerve(s), suggesting that a very long peripheral nerve block-lasting many months rather than hours-may permanently reverse the abnormal changes in the brain, and provide definitive relief from phantom pain. A prolonged nerve block lasting a few months may be provided by freezing the nerve using a process called "cryoneurolysis". The ultimate objective of the proposed research study is to determine if cryoanalgesia is an effective treatment for intractable post-amputation phantom limb pain. The proposed research study will include subjects with an existing lower extremity amputation who experience intractable daily phantom limb pain. A single ultrasound-guided treatment of cryoneurolysis (or sham block-determined randomly like a flip of a coin) will be applied to the target nerve(s) involved with the phantom pain. Although not required, each subject may return four months later for the alternative treatment (if the first treatment is sham, then the second treatment would be cryoneurolysis) so that all participants have the option of receiving the active treatment. Subjects will be followed for a total of 12 months with data collected by telephone.

DETAILED DESCRIPTION:
Subjects will be asked to make no changes to their analgesic regimen for at least 1 month prior to the cryoneurolysis procedure and continuing for 4 months until the measurement of the primary end point-for the duration of the study, all patients will be allowed to continue their pre-intervention analgesics. All subjects will have a peripheral intravenous catheter inserted, standard noninvasive monitors applied, and oxygen administered via a facemask or nasal cannula. Midazolam and fentanyl (IV) will be titrated for patient comfort. The specific nerves targeted will be the sciatic and femoral (or their distal branches). The potential cryoneurolysis sites will be cleansed with chlorhexidine gluconate and isopropyl alcohol. The target nerves will be identified in a transverse cross-sectional (short axis) view using ultrasound. A Tuohy-tip needle will be inserted beneath the ultrasound transducer and directed until the needle tip is immediately adjacent to the target nerve. Local anesthetic (1-3 mL, lidocaine 2%) will be injected. This will be repeated for the femoral nerve. Within 20 minutes of the second injection, the subject's limb pain level will be evaluated on the 0-10 NRS and if higher than at baseline prior to injection, the subject will NOT continue with treatment and their participation in the study will terminate upon discharge.

Treatment group assignment (randomization). Remaining subjects will be allocated to one of two possible treatments:

1. cryoneurolysis
2. sham cryoneurolysis (placebo control)

Randomization will be computer-generated and stratified by enrolling institution in randomly chosen block sizes. Cryoneurolysis probes are available that either (1) pass nitrous oxide to the tip inducing freezing temperatures; or, (2) vent the nitrous oxide at the base of the probe so that no gas reaches the probe tip, resulting in no temperature change (PainBlocker, Epimed, Farmers Branch, Texas). Importantly, these probes are indistinguishable in appearance. Unmasking will not occur until statistical analysis is complete.

Intervention. The potential cryoneurolysis sites will be again cleansed with chlorhexidine gluconate and isopropyl alcohol. With the same ultrasound transducer used to previously administer local anesthetic, the target nerve will again be identified in a transverse cross-sectional (short axis) view at or distal to the deposition of local anesthetic. A cryoneurolysis device (PainBlocker, Epimed, Farmers Branch, Texas) will be inserted with the appropriate randomization-designated probe (either active or sham/placebo) and nitrous oxide. The cryoneurolysis device will be triggered using 3 cycles of 2-minute gas activation (active or sham) separated by 1-minute defrost periods. The process will be repeated with the same treatment probe for the femoral nerve (e.g., both nerves will receive either active cryoneurolysis or sham/placebo, and not a mix of the two possible treatments).

Optional crossover treatment. Four to 6 months following the initial treatment, subjects may return for an optional repeated intervention procedure ("crossover") with the alternative treatment (either active cryoneurolysis or sham/placebo), again in a double-masked fashion using the same protocol as described for the initial intervention. The crossover treatment is not required for study participation, as the primary analyses will include a parallel study design for the initial intervention evaluated prior to any crossover treatment. This crossover will not affect the primary analyses, which will involve a parallel group study design and investigate the effects of cryoneurolysis within 4 months of the initial intervention.

Outcome measurements (endpoints). The primary end point will be the difference in average daily phantom pain intensity at baseline and 4 months following the initial intervention (measured with the NRS as part of the Brief Pain Inventory). The primary analyses will compare the two treatments (inter-subject comparisons) during the initial treatment period in which half of the subjects will receive active cryoneurolysis and the other half a sham/placebo treatment. Endpoints will be evaluated at baseline and post-treatment (Day 0), Days 1 and 7; and Months 1, 2, 3, 4, and 12. These same time points through Month 4 will be evaluated following the optional second (crossover) treatment.

Data collection. The questionnaires for all subjects-regardless of enrolling center-will be administered by telephone from the University of California San Diego by research coordinators specifically trained in these instruments' application, minimizing inter-rater discordance. Staff masked to treatment group assignment will perform all assessments.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of at least 18 years of age
* with a lower limb traumatic or surgical amputation at least 12 weeks prior to enrollment distal to the hip (femoral head remaining)
* who experience at least moderate phantom limb pain-defined as a 3 or higher on the Numeric Rating Scale (NRS; 0-10, 0= no pain; 10=worst imaginable pain)-at least daily for the previous 2 months.
* accepting of a cryoneurolysis procedure
* willing to avoid both changes to their analgesic regimen as well as elective surgical procedures from 1 month prior to and at least 4 months following the initial cryoneurolysis procedure.

Exclusion Criteria:

* allergy to amide local anesthetics
* pregnancy
* incarceration
* inability to communicate with the investigators
* morbid obesity (body mass index > 40 kg/m2)
* possessing any contraindication specific to cryoneurolysis such as a localized infection at the treatment site, cryoglobulinemia, cold urticaria and Reynaud's Syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2018-03-23 (Actual); Primary Completion 2021-08-17 (Actual); Study Completion 2022-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Ilfeld, MD, MS, Principal Investigator — University California San Diego Department of Anesthesiology; Rodney Gabriel, MD, MAS, Study Director — University California San Diego Department of Anesthesiology
Locations (6):
- United States (6):
  - Veterans Affairs Palo Alto Health Care System, Palo Alto, California
  - University California San Diego, San Diego, California
  - Naval Medical Center San Diego (NMCSD), San Diego, California
  - University of Florida, Gainesville, Florida
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Undecided
Pending

REFERENCES:
- [Result] Moesker AA, Karl HW, Trescot AM. Treatment of phantom limb pain by cryoneurolysis of the amputated nerve. Pain Pract. 2014 Jan;14(1):52-6. doi: 10.1111/papr.12020. Epub 2012 Dec 19. PMID 23279331

RESULTS

PARTICIPANT FLOW:
Groups:
- Cryoneurolysis, Then Optional Crossover Sham: Cryoneurolysis of the femoral and sciatic nerves (or their distal counterparts) in the residual limb: The cryoneurolysis device will be triggered using 3 cycles of 2-minute gas activation separated by 1-minute defrost periods. For active probes, the nitrous oxide will be deployed to the tip where a drop in temperature to -70°C will result in cryoneurolysis.
  Cryoneurolysis: Cryoneurolysis of the femoral and sciatic nerves (or their distal counterparts) in the residual limb: The cryoneurolysis device will be triggered using 3 cycles of 2-minute gas activation separated by 1-minute defrost periods. For active probes, the nitrous oxide will be deployed to the tip where a drop in temperature to -70°C will result in cryoneurolysis.
  Optional crossover: Sham cryoneurolysis of the femoral and sciatic nerves (or their distal counterparts) in the residual limb: The cryoneurolysis device will be triggered using 3 cycles of 2-minute gas activation separated by 1-minute defrost periods. However, for sham probes, the nitrous oxide is not deployed to the tip and therefore there is no drop in temperature resulting in cryoneurolysis.
- Sham, Then Optional Crossover Cryoneurolysis: Sham cryoneurolysis of the femoral and sciatic nerves (or their distal counterparts) in the residual limb: The cryoneurolysis device will be triggered using 3 cycles of 2-minute gas activation separated by 1-minute defrost periods. However, for sham probes, the nitrous oxide is not deployed to the tip and therefore there is no drop in temperature resulting in cryoneurolysis.
  Sham Comparator: Sham cryoneurolysis of the femoral and sciatic nerves (or their distal counterparts) in the residual limb: The cryoneurolysis device will be triggered using 3 cycles of 2-minute gas activation separated by 1-minute defrost periods. However, for sham probes, the nitrous oxide is not deployed to the tip and therefore there is no drop in temperature resulting in cryoneurolysis.
  Optional crossover: Cryoneurolysis of the femoral and sciatic nerves (or their distal counterparts) in the residual limb: The cryoneurolysis device will be triggered using 3 cycles of 2-minute gas activation separated by 1-minute defrost periods. For active probes, the nitrous oxide will be deployed to the tip where a drop in temperature to -70°C will result in cryoneurolysis.
Period: Initial Treatment
Arm/Group | Cryoneurolysis, Then Optional Crossover Sham | Sham, Then Optional Crossover Cryoneurolysis
Started | 71 | 73
Completed | 71 | 73
Not Completed | 0 | 0
Period: Optional Crossover Treatment
Arm/Group | Cryoneurolysis, Then Optional Crossover Sham | Sham, Then Optional Crossover Cryoneurolysis
Started | 71 | 73
Completed | 42 | 49
Not Completed | 29 | 24

BASELINE CHARACTERISTICS:
Groups:
- Cryoneurolysis, Then Optional Crossover Sham: Cryoneurolysis of the femoral and sciatic nerves (or their distal counterparts) in the residual limb: The cryoneurolysis device will be triggered using 3 cycles of 2-minute gas activation separated by 1-minute defrost periods. For active probes, the nitrous oxide will be deployed to the tip where a drop in temperature to -70°C will result in cryoneurolysis.
  Cryoneurolysis: Cryoneurolysis of the femoral and sciatic nerves (or their distal counterparts) in the residual limb: The cryoneurolysis device will be triggered using 3 cycles of 2-minute gas activation separated by 1-minute defrost periods. For active probes, the nitrous oxide will be deployed to the tip where a drop in temperature to -70°C will result in cryoneurolysis.
- Sham, Then Optional Crossover Cryoneurolysis: Sham cryoneurolysis of the femoral and sciatic nerves (or their distal counterparts) in the residual limb: The cryoneurolysis device will be triggered using 3 cycles of 2-minute gas activation separated by 1-minute defrost periods. However, for sham probes, the nitrous oxide is not deployed to the tip and therefore there is no drop in temperature resulting in cryoneurolysis.
  Sham Comparator: Sham cryoneurolysis of the femoral and sciatic nerves (or their distal counterparts) in the residual limb: The cryoneurolysis device will be triggered using 3 cycles of 2-minute gas activation separated by 1-minute defrost periods. However, for sham probes, the nitrous oxide is not deployed to the tip and therefore there is no drop in temperature resulting in cryoneurolysis.
- Total: Total of all reporting groups
Arm/Group | Cryoneurolysis, Then Optional Crossover Sham | Sham, Then Optional Crossover Cryoneurolysis | Total
Number analyzed (Participants) | 71 | 73 | 144
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (13) | 58 (13) | 58 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 29 | 47
  Male | 53 | 44 | 97
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 71 | 73 | 144
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 29 (5.8) | 28 (5.3) | 28 (5.5)
Marital status [Count of Participants; unit: Participants]
  Single (never married) | 16 | 16 | 32
  Single (divorced) | 18 | 12 | 30
  Currently married | 33 | 36 | 69
  Others (separated or widowed) | 4 | 9 | 13
Military Status [Count of Participants; unit: Participants]
  Civilian (never in military) | 59 | 55 | 114
  Veteran | 11 | 18 | 29
  Active Duty | 1 | 0 | 1
Years of education [Median (Inter-Quartile Range); unit: years] | 14 [12 to 16] | 14 [12 to 16] | 14 [12 to 16]
Amputation Information [Count of Participants; unit: Participants]
  Trans-femoral | 22 | 21 | 43
  Trans-tibial | 46 | 46 | 92
  Foot/ankle | 3 | 6 | 9
History of residual limb pain [Count of Participants; unit: Participants] | 55 | 55 | 110
Current residual limb pain [Count of Participants; unit: Participants] | 44 | 45 | 89
Current prosthesis use [Count of Participants; unit: Participants] | 66 | 67 | 133
Distance of treatment from end of residual limb [Median (Inter-Quartile Range); unit: cm]
  Sciatic nerve | 15 [11 to 23] | 17 [12 to 23] | 16 [11 to 23]
  Femoral nerve | 22 [15 to 31] | 22 [16 to 33] | 22 [15 to 32]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average Daily Phantom Pain Intensity
Description: The difference in average daily phantom pain intensity at baseline and 4 months following the initial intervention (measured with the numeric rating scale as part of the Brief Pain Inventory with a minimum value of 0 and maximum value of 10, 0=no pain and 10=worst imaginable pain)
Time Frame: Baseline and 4 months later (difference between the two is the primary end point)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Cryoneurolysis, Then Optional Crossover Sham: Initial treatment: Cryoneurolysis of the femoral and sciatic nerves (or their distal counterparts) in the residual limb: The cryoneurolysis device will be triggered using 3 cycles of 2-minute gas activation separated by 1-minute defrost periods. For active probes, the nitrous oxide will be deployed to the tip where a drop in temperature to -70°C will result in cryoneurolysis.
  Crossover treatment: Sham cryoneurolysis of the femoral and sciatic nerves (or their distal counterparts) in the residual limb: The cryoneurolysis device will be triggered using 3 cycles of 2-minute gas activation separated by 1-minute defrost periods. However, for sham probes, the nitrous oxide is not deployed to the tip and therefore there is no drop in temperature resulting in cryoneurolysis.
- Sham, Then Optional Crossover Cryoneurolysis: Initial treatment: Sham cryoneurolysis of the femoral and sciatic nerves (or their distal counterparts) in the residual limb: The cryoneurolysis device will be triggered using 3 cycles of 2-minute gas activation separated by 1-minute defrost periods. However, for sham probes, the nitrous oxide is not deployed to the tip and therefore there is no drop in temperature resulting in cryoneurolysis.
  Crossover treatment: Cryoneurolysis of the femoral and sciatic nerves (or their distal counterparts) in the residual limb: The cryoneurolysis device will be triggered using 3 cycles of 2-minute gas activation separated by 1-minute defrost periods. For active probes, the nitrous oxide will be deployed to the tip where a drop in temperature to -70°C will result in cryoneurolysis.
Arm/Group | Cryoneurolysis, Then Optional Crossover Sham | Sham, Then Optional Crossover Cryoneurolysis
Number analyzed (Participants) | 71 | 73
score on a scale | 0.5 [-0.5 to 3.0] | 0 [0 to 3]

2. Secondary Outcome: Average Daily Phantom Pain Intensity
Description: The average daily phantom pain intensity at between 1 day and 12 months following the initial intervention (measured with the numeric rating scale as part of the Brief Pain Inventory with a minimum value of 0 and maximum value of 10, 0=no pain and 10=worst imaginable pain)
  To read the results: for the group that received cryoneurolysis initially followed by sham for the crossover treatment, "initial" Days 1 - Month 4 provide the results for those receiving cryoneurolysis while "crossover" Days 1 - Month 4 provide the results for those receiving sham treatment. This is reversed for the other treatment group that received sham initially followed by cryoneurolysis for the crossover treatment.
Time Frame: Endpoints will be evaluated at baseline and on Days 1 and 7; and Months 1, 2, 3, and 4 after both the initial and subsequently the crossover treatments; and 12 months after the initial treatment
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Cryoneurolysis Initial Treatment, Sham Crossover Treatment: Initial treatment: Cryoneurolysis of the femoral and sciatic nerves (or their distal counterparts) in the residual limb: The cryoneurolysis device will be triggered using 3 cycles of 2-minute gas activation separated by 1-minute defrost periods. For active probes, the nitrous oxide will be deployed to the tip where a drop in temperature to -70°C will result in cryoneurolysis.
  Crossover treatment: Sham cryoneurolysis of the femoral and sciatic nerves (or their distal counterparts) in the residual limb: The cryoneurolysis device will be triggered using 3 cycles of 2-minute gas activation separated by 1-minute defrost periods. However, for sham probes, the nitrous oxide is not deployed to the tip and therefore there is no drop in temperature resulting in cryoneurolysis.
- Sham Comparator Initial Treatment, Cryoneurolysis Crossover Treatment: Initial treatment: Sham cryoneurolysis of the femoral and sciatic nerves (or their distal counterparts) in the residual limb: The cryoneurolysis device will be triggered using 3 cycles of 2-minute gas activation separated by 1-minute defrost periods. However, for sham probes, the nitrous oxide is not deployed to the tip and therefore there is no drop in temperature resulting in cryoneurolysis.
  Crossover treatment: Cryoneurolysis of the femoral and sciatic nerves (or their distal counterparts) in the residual limb: The cryoneurolysis device will be triggered using 3 cycles of 2-minute gas activation separated by 1-minute defrost periods. For active probes, the nitrous oxide will be deployed to the tip where a drop in temperature to -70°C will result in cryoneurolysis.
Arm/Group | Cryoneurolysis Initial Treatment, Sham Crossover Treatment | Sham Comparator Initial Treatment, Cryoneurolysis Crossover Treatment
Number analyzed (Participants) | 71 | 73
score on a scale
  Day 0 (baseline) | 5 [4 to 6] | 5 [4 to 7]
  Day 1, initial treatment | 0 [0 to 4] | 1 [0 to 5]
  Day 7, initial treatment | 3 [0 to 5] | 3.5 [0 to 5]
  Month 1, initial treatment | 3.5 [0 to 5] | 4 [0 to 6]
  Month 2, initial treatment | 3 [0 to 5] | 4 [2 to 5]
  Month 3, initial treatment | 3.5 [0 to 5] | 5 [2 to 6]
  Month 4, initial treatment | 4.3 [1.5 to 6] | 4.5 [2 to 6]
  Day 0, crossover treatment | 5 [3 to 7] | 5 [4 to 6]
  Day 1, crossover treatment | 0 [0 to 3] | 0 [0 to 2.5]
  Day 7, crossover treatment | 0 [0 to 2] | 0 [0 to 5]
  Month 1, crossover treatment | 2 [0 to 4] | 3 [0 to 5]
  Month 2, crossover treatment | 2 [0 to 4] | 3 [0 to 5]
  Month 3, crossover treatment | 2 [0 to 4] | 3 [0 to 5]
  Month 4, crossover treatment | 2 [0 to 4] | 3.5 [0 to 5]
  Month 12, initial | 1 [0 to 4] | 3 [0 to 5]

3. Secondary Outcome: Worst Daily Phantom Pain Intensity
Description: The worst daily phantom pain intensity at between 1 day and 12 months following the initial intervention (measured with the numeric rating scale as part of the Brief Pain Inventory with a minimum value of 0 and maximum value of 10, 0=no pain and 10=worst imaginable pain). The worst pain is the maximum experienced in the previous 72 hour period (except day 1 which is the previous 24 hour period).
  To read the results: for the group that received cryoneurolysis initially followed by sham for the crossover treatment, "initial" Days 1 - Month 4 provide the results for those receiving cryoneurolysis while "crossover" Days 1 - Month 4 provide the results for those receiving sham treatment. This is reversed for the other treatment group that received sham initially followed by cryoneurolysis for the crossover treatment.
Time Frame: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Cryoneurolysis Initial, Sham Crossover: Initial treatment: Cryoneurolysis of the femoral and sciatic nerves (or their distal counterparts) in the residual limb: The cryoneurolysis device will be triggered using 3 cycles of 2-minute gas activation separated by 1-minute defrost periods. For active probes, the nitrous oxide will be deployed to the tip where a drop in temperature to -70°C will result in cryoneurolysis.
  Crossover treatment: Sham cryoneurolysis of the femoral and sciatic nerves (or their distal counterparts) in the residual limb: The cryoneurolysis device will be triggered using 3 cycles of 2-minute gas activation separated by 1-minute defrost periods. However, for sham probes, the nitrous oxide is not deployed to the tip and therefore there is no drop in temperature resulting in cryoneurolysis.
- Sham Comparator Initial, Cryoneurolysis Crossover: Initial treatment: Sham cryoneurolysis of the femoral and sciatic nerves (or their distal counterparts) in the residual limb: The cryoneurolysis device will be triggered using 3 cycles of 2-minute gas activation separated by 1-minute defrost periods. However, for sham probes, the nitrous oxide is not deployed to the tip and therefore there is no drop in temperature resulting in cryoneurolysis.
  Crossover treatment: Cryoneurolysis of the femoral and sciatic nerves (or their distal counterparts) in the residual limb: The cryoneurolysis device will be triggered using 3 cycles of 2-minute gas activation separated by 1-minute defrost periods. For active probes, the nitrous oxide will be deployed to the tip where a drop in temperature to -70°C will result in cryoneurolysis.
Arm/Group | Cryoneurolysis Initial, Sham Crossover | Sham Comparator Initial, Cryoneurolysis Crossover
Number analyzed (Participants) | 71 | 73
score on a scale
  Day 0 (baseline) | 8 [7 to 9] | 8 [7 to 10]
  Day 1, initial treatment | 2.5 [0 to 7] | 3 [0 to 7]
  Day 7, initial treatment | 6 [0 to 8.5] | 6 [0 to 9]
  Month 1, initial treatment | 6.5 [0 to 9] | 7 [0 to 9]
  Month 2, initial treatment | 7 [1 to 9] | 7 [4 to 9]
  Month 3, initial treatment | 7 [2 to 9] | 8 [5 to 9]
  Month 4, initial treatment | 7.5 [4 to 9] | 8 [5 to 9]
  Day 0, crossover treatment | 8 [6.5 to 9.5] | 8 [6 to 9]
  Day 1, crossover treatment | 0 [0 to 5] | 0 [0 to 6]
  Day 7, crossover treatment | 0 [0 to 7] | 5.25 [0 to 8.5]
  Month 1, crossover treatment | 5 [0 to 8] | 6 [1 to 8]
  Month 2, crossover treatment | 6 [0 to 7] | 6 [3 to 7.5]
  Month 3, crossover treatment | 6 [0 to 8] | 7 [4 to 8]
  Month 4, crossover treatment | 6 [0 to 8] | 6.5 [3 to 8]
  Month 12, initial | 6 [0 to 9] | 7 [3 to 8]

4. Secondary Outcome: Residual Limb Pain, Average
Description: Residual limb pain will be assessed using a Numeric Rating Scale which is a highly-sensitive measure of pain intensity with numbers ranging from 0 to 10, with zero equivalent to no pain and 10 equivalent to the worst imaginable pain.
  To read the results: for the group that received cryoneurolysis initially followed by sham for the crossover treatment, "initial" Days 1 - Month 4 provide the results for those receiving cryoneurolysis while "crossover" Days 1 - Month 4 provide the results for those receiving sham treatment. This is reversed for the other treatment group that received sham initially followed by cryoneurolysis for the crossover treatment.
Time Frame: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Cryoneurolysis, Then Optional Crossover Sham | Sham, Then Optional Crossover Cryoneurolysis
Number analyzed (Participants) | 71 | 73
score on a scale
  Day 0 (baseline) | 3 [0 to 6] | 3 [0 to 5]
  Day 1, initial treatment | 0 [0 to 1] | 0 [0 to 2]
  Day 7, initial treatment | 0 [0 to 4] | 0 [0 to 3.5]
  Month 1, initial treatment | 0 [0 to 4] | 0 [0 to 3.5]
  Month 2, initial treatment | 0 [0 to 3.5] | 0 [0 to 4]
  Month 3, initial treatment | 0 [0 to 4] | 0 [0 to 4]
  Month 4, initial treatment | 0.5 [0 to 4] | 0.5 [0 to 4.5]
  Day 0, crossover treatment | 3 [.25 to 5] | 3 [0 to 6]
  Day 1, crossover treatment | 0 [0 to 1] | 0 [0 to 0]
  Day 7, crossover treatment | 0 [0 to 2] | 0 [0 to 3]
  Month 1, crossover treatment | 0 [0 to 4] | 2 [0 to 4]
  Month 2, crossover treatment | 0 [0 to 2.5] | 0 [0 to 4]
  Month 3, crossover treatment | 0 [0 to 1] | 0 [0 to 5]
  Month 4, crossover treatment | 0 [0 to 3] | 0 [0 to 4]
  Month 12, initial | 0 [0 to 1] | 0 [0 to 3]

5. Secondary Outcome: Residual Limb Pain, Worst
Description: Residual limb pain will be assessed using a Numeric Rating Scale which is a highly-sensitive measure of pain intensity with numbers ranging from 0 to 10, with zero equivalent to no pain and 10 equivalent to the worst imaginable pain. The worst pain is the maximum experienced over the previous 72 hours (24 hours for Day 1).
  To read the results: for the group that received cryoneurolysis initially followed by sham for the crossover treatment, "initial" Days 1 - Month 4 provide the results for those receiving cryoneurolysis while "crossover" Days 1 - Month 4 provide the results for those receiving sham treatment. This is reversed for the other treatment group that received sham initially followed by cryoneurolysis for the crossover treatment.
Time Frame: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Sham Comparator Initially, Cryoneurolysis Crossover: Initial treatment: Sham cryoneurolysis of the femoral and sciatic nerves (or their distal counterparts) in the residual limb: The cryoneurolysis device will be triggered using 3 cycles of 2-minute gas activation separated by 1-minute defrost periods. However, for sham probes, the nitrous oxide is not deployed to the tip and therefore there is no drop in temperature resulting in cryoneurolysis.
  Crossover treatment: Cryoneurolysis of the femoral and sciatic nerves (or their distal counterparts) in the residual limb: The cryoneurolysis device will be triggered using 3 cycles of 2-minute gas activation separated by 1-minute defrost periods. For active probes, the nitrous oxide will be deployed to the tip where a drop in temperature to -70°C will result in cryoneurolysis.
Arm/Group | Cryoneurolysis, Then Optional Crossover Sham | Sham Comparator Initially, Cryoneurolysis Crossover
Number analyzed (Participants) | 71 | 73
score on a scale
  Day 0 (baseline) | 6 [0 to 8] | 5 [0 to 8]
  Day 1, initial treatment | 0 [0 to 5] | 0 [0 to 5]
  Day 7, initial treatment | 0 [0 to 6] | 0 [0 to 6]
  Month 1, initial treatment | 0 [0 to 7] | 1 [0 to 6.5]
  Month 2, initial treatment | 0 [0 to 6] | 0 [0 to 7]
  Month 3, initial treatment | 0 [0 to 7] | 0 [0 to 7]
  Month 4, initial treatment | 3 [0 to 8] | 2 [0 to 8]
  Day 0, crossover treatment | 6.5 [3 to 8] | 6 [0 to 8]
  Day 1, crossover treatment | 0 [0 to 2] | 0 [0 to 1.5]
  Day 7, crossover treatment | 0 [0 to 6] | 1.25 [0 to 7]
  Month 1, crossover treatment | 0 [0 to 8] | 5 [0 to 8]
  Month 2, crossover treatment | 0 [0 to 5.5] | 0 [0 to 7]
  Month 3, crossover treatment | 0 [0 to 6] | 0 [0 to 6]
  Month 4, crossover treatment | 0 [0 to 7] | 2 [0 to 8]
  Month 12, initial | 0 [0 to 6] | 0 [0 to 7]

6. Secondary Outcome: Patient Global Impression of Change
Description: The Patient Global Impression of Change Scale is a 7-point ordinal scale requiring the subject to rate the current severity of their global situation as it relates to phantom limb pain (as defined by each individual) compared to their baseline. This scale has the words "very much worse" to the left by the number one, and "very much improved" to the right, adjacent to the number seven. The words "no change" are in the middle of the scale above the number four. The Patient Global Impression of Change Scale has been validated in over ten prospective trials, including studies specifically involving peripheral neuropathy
  To read the results: for the group that received cryoneurolysis initially followed by sham for the crossover treatment, "initial" Days 1 - Month 4 provide the results for those receiving cryoneurolysis while "crossover" Days 1 - Month 4 provide the results for those receiving sham treatment. This is reversed for the other treatment group that received sham initially f
Time Frame: Endpoints will be evaluated on Days 1 and 7; and Months 1, 2, 3, and 4 after both the initial and subsequently the crossover treatments; and 12 months after the initial treatment
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Sham Comparator Initially, Cryoneurolysis Crossover Treatment: Initial treatment: Cryoneurolysis of the femoral and sciatic nerves (or their distal counterparts) in the residual limb: The cryoneurolysis device will be triggered using 3 cycles of 2-minute gas activation separated by 1-minute defrost periods. For active probes, the nitrous oxide will be deployed to the tip where a drop in temperature to -70°C will result in cryoneurolysis.
  Crossover treatment: Sham cryoneurolysis of the femoral and sciatic nerves (or their distal counterparts) in the residual limb: The cryoneurolysis device will be triggered using 3 cycles of 2-minute gas activation separated by 1-minute defrost periods. However, for sham probes, the nitrous oxide is not deployed to the tip and therefore there is no drop in temperature resulting in cryoneurolysis.
Arm/Group | Cryoneurolysis Initial Treatment, Sham Crossover Treatment | Sham Comparator Initially, Cryoneurolysis Crossover Treatment
Number analyzed (Participants) | 71 | 73
score on a scale
  Day 1, initial treatment | 7 [4 to 7] | 6 [4 to 7]
  Day 7, initial treatment | 5 [4 to 7] | 4 [4 to 7]
  Month 1, initial treatment | 4 [4 to 7] | 4 [4 to 7]
  Month 2, initial treatment | 4 [4 to 7] | 4 [4 to 6]
  Month 3, initial treatment | 4 [4 to 7] | 4 [4 to 5]
  Month 4, initial treatment | 4 [4 to 7] | 4 [4 to 6]
  Day 1, crossover treatment | 7 [6 to 7] | 7 [5 to 7]
  Day 7, crossover treatment | 7 [6 to 7] | 6 [4 to 7]
  Month 1, crossover treatment | 6 [4 to 7] | 4 [4 to 7]
  Month 2, crossover treatment | 6 [4 to 7] | 5 [4 to 7]
  Month 3, crossover treatment | 6 [4 to 7] | 4 [4 to 7]
  Month 4, crossover treatment | 6 [4 to 7] | 4 [4 to 7]
  Month 12, initial | 6 [4 to 7] | 5 [4 to 7]

7. Secondary Outcome: Brief Pain Inventory Interference Subscale
Description: The Brief Pain Inventory (interference sub scale) is an instrument that measures the interference with physical and emotional functioning using a 0-10 scale (0 = no interference; 10 = complete interference). The seven interference questions involve general activity, mood, walking ability, normal work activities (both inside and outside of the home), relationships, sleep, and enjoyment of life. The seven functioning questions can be added to produce an interference subscale (0-70). A higher score reveals more interference with physical and emotional functioning.
  To read the results: for the group that received cryoneurolysis initially followed by sham for the crossover treatment, "initial" Days 1 - Month 4 provide the results for those receiving cryoneurolysis while "crossover" Days 1 - Month 4 provide the results for those receiving sham treatment. This is reversed for the other treatment group that received sham initially followed by cryoneurolysis for the crossover treatment.
Time Frame: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Sham Comparator Initially, Cryoneurolysis Crossover Treatment: Initial treatment: Sham cryoneurolysis of the femoral and sciatic nerves (or their distal counterparts) in the residual limb: The cryoneurolysis device will be triggered using 3 cycles of 2-minute gas activation separated by 1-minute defrost periods. However, for sham probes, the nitrous oxide is not deployed to the tip and therefore there is no drop in temperature resulting in cryoneurolysis.
  Crossover treatment: Cryoneurolysis of the femoral and sciatic nerves (or their distal counterparts) in the residual limb: The cryoneurolysis device will be triggered using 3 cycles of 2-minute gas activation separated by 1-minute defrost periods. For active probes, the nitrous oxide will be deployed to the tip where a drop in temperature to -70°C will result in cryoneurolysis.
Arm/Group | Cryoneurolysis Initial Treatment, Sham Crossover Treatment | Sham Comparator Initially, Cryoneurolysis Crossover Treatment
Number analyzed (Participants) | 71 | 73
score on a scale
  Day 0 (baseline) | 36 [21 to 47] | 34 [22 to 43]
  Day 1, initial treatment | 0 [0 to 22] | 0 [0 to 19]
  Day 7, initial treatment | 7 [0 to 32] | 19 [0 to 34]
  Month 1, initial treatment | 15 [0 to 40] | 22 [2 to 33]
  Month 2, initial treatment | 10 [0 to 40] | 22 [2 to 35]
  Month 3, initial treatment | 13 [0 to 38] | 21 [5 to 38]
  Month 4, initial treatment | 20 [0 to 38] | 19 [4 to 32]
  Day 0, crossover treatment | 26 [10 to 42] | 27 [20 to 39]
  Day 1, crossover treatment | 0 [0 to 7] | 0 [0 to 7]
  Day 7, crossover treatment | 0 [0 to 14] | 2 [0 to 32]
  Month 1, crossover treatment | 4 [0 to 28] | 12 [0 to 31]
  Month 2, crossover treatment | 10 [0 to 21.5] | 14 [0 to 35]
  Month 3, crossover treatment | 9 [0 to 22] | 18 [0 to 31]
  Month 4, crossover treatment | 11 [0 to 24] | 17 [0 to 34]
  Month 12, initial | 14 [4 to 33] | 12 [2 to 35]

8. Secondary Outcome: Beck Depression Inventory
Description: The Beck Depression Inventory is a 21-item instrument that measures characteristic symptoms and signs of depression, requires only a 5th grade comprehension level to adequately understand the questions, and demonstrates a high internal consistency (0.73-0.92, mean of 0.86), reliability and validity. Each of the 21 factors is rated on a 0-3 scale, and then summed to produce the total score of 0-63. Mild, moderate, and severe depression is defined with scores of 10-18, 19-29, and 30-63, respectively.
  To read the results: for the group that received cryoneurolysis initially followed by sham for the crossover treatment, "initial" Month 4 provides the results for those receiving cryoneurolysis while "crossover" Month 4 provides the results for those receiving sham treatment. This is reversed for the other treatment group that received sham initially followed by cryoneurolysis for the crossover treatment.
Time Frame: At baseline, 4 months after the initial and crossover treatments as well as 12 months after the initial treatment
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Cryoneurolysis Initial Treatment, Sham Crossover Treatment | Sham Comparator Initially, Cryoneurolysis Crossover Treatment
Number analyzed (Participants) | 71 | 73
score on a scale
  Baseline (Day 0) | 10 [5 to 17] | 9 [4 to 13]
  Month 4, initial treatment | 4 [0 to 14] | 2 [0 to 9]
  Month 4, crossover treatment | 0 [0 to 5] | 0 [0 to 6]
  Month 12, initial | 0 [0 to 7] | 0 [0 to 3]

9. Secondary Outcome: Phantom Limb Pain Frequency
Description: Pain perceived to emanate from part of the injured limb that no longer exists. The frequency is the number of times this is experienced in the previous 72 hours.
  To read the results: for the group that received cryoneurolysis initially followed by sham for the crossover treatment, "initial" Days 1 - Month 4 provide the results for those receiving cryoneurolysis while "crossover" Days 1 - Month 4 provide the results for those receiving sham treatment. This is reversed for the other treatment group that received sham initially followed by cryoneurolysis for the crossover treatment.
Time Frame: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Occurrences
Arm/Group | Cryoneurolysis Initial Treatment, Sham Crossover Treatment | Sham Comparator Initially, Cryoneurolysis Crossover Treatment
Number analyzed (Participants) | 71 | 73
Occurrences
  Baseline (Day 0) | 24 [12 to 24] | 24 [16 to 24]
  Day 1, initial treatment | 1 [0 to 24] | 2 [0 to 24]
  Day 7, initial treatment | 9 [0 to 24] | 24 [2 to 24]
  Month 1, initial treatment | 11 [1 to 24] | 24 [1 to 24]
  Month 2, initial treatment | 15 [1 to 24] | 24 [3 to 24]
  Month 3, initial treatment | 24 [1 to 24] | 24 [5 to 24]
  Month 4, initial treatment | 24 [2 to 24] | 24 [4 to 24]
  Day 0, crossover treatment | 22 [4 to 24] | 24 [5 to 24]
  Day 1, crossover treatment | 0 [0 to 24] | 0 [0 to 24]
  Day 7, crossover treatment | 0 [0 to 20] | 4.5 [0 to 24]
  Month 1, crossover treatment | 4 [0 to 24] | 12 [1 to 24]
  Month 2, crossover treatment | 3 [0 to 24] | 15 [1 to 24]
  Month 3, crossover treatment | 7.5 [0 to 24] | 9 [3 to 24]
  Month 4, crossover treatment | 8 [0 to 24] | 24 [2 to 24]
  Month 12, initial | 3 [0 to 24] | 4 [1 to 24]

10. Secondary Outcome: Phantom Limb Pain Duration
Description: Pain perceived to emanate from part of the injured limb that no longer exists. The duration is the average number of hours that each occurrence is experienced in the previous 72 hours.
  To read the results: for the group that received cryoneurolysis initially followed by sham for the crossover treatment, "initial" Days 1 - Month 4 provide the results for those receiving cryoneurolysis while "crossover" Days 1 - Month 4 provide the results for those receiving sham treatment. This is reversed for the other treatment group that received sham initially followed by cryoneurolysis for the crossover treatment.
Time Frame: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: hours
Groups:
- Cryoneurolysis Initial Treatment; Sham Crossover Treatment: Initial treatment: Cryoneurolysis of the femoral and sciatic nerves (or their distal counterparts) in the residual limb: The cryoneurolysis device will be triggered using 3 cycles of 2-minute gas activation separated by 1-minute defrost periods. For active probes, the nitrous oxide will be deployed to the tip where a drop in temperature to -70°C will result in cryoneurolysis.
  Crossover treatment: Sham cryoneurolysis of the femoral and sciatic nerves (or their distal counterparts) in the residual limb: The cryoneurolysis device will be triggered using 3 cycles of 2-minute gas activation separated by 1-minute defrost periods. However, for sham probes, the nitrous oxide is not deployed to the tip and therefore there is no drop in temperature resulting in cryoneurolysis.
- Sham Comparator Initially, Cryoneuorlysis Crossover Treatment: Initial treatment: Sham cryoneurolysis of the femoral and sciatic nerves (or their distal counterparts) in the residual limb: The cryoneurolysis device will be triggered using 3 cycles of 2-minute gas activation separated by 1-minute defrost periods. However, for sham probes, the nitrous oxide is not deployed to the tip and therefore there is no drop in temperature resulting in cryoneurolysis.
  Crossover treatment: Cryoneurolysis of the femoral and sciatic nerves (or their distal counterparts) in the residual limb: The cryoneurolysis device will be triggered using 3 cycles of 2-minute gas activation separated by 1-minute defrost periods. For active probes, the nitrous oxide will be deployed to the tip where a drop in temperature to -70°C will result in cryoneurolysis.
Arm/Group | Cryoneurolysis Initial Treatment; Sham Crossover Treatment | Sham Comparator Initially, Cryoneuorlysis Crossover Treatment
Number analyzed (Participants) | 71 | 73
hours
  Baseline (Day 0) | 24 [1 to 24] | 24 [2 to 24]
  Day 1, initial treatment | 0 [0 to 24] | 0 [0 to 24]
  Day 7, initial treatment | 0 [0 to 24] | 3 [0 to 24]
  Month 1, initial treatment | 1 [0 to 24] | 2 [0 to 24]
  Month 2, initial treatment | 2 [0 to 24] | 24 [0 to 24]
  Month 3, initial treatment | 24 [0 to 24] | 24 [0 to 24]
  Month 4, initial treatment | 15 [0 to 24] | 24 [0 to 24]
  Day 0, crossover treatment | 13.5 [0 to 24] | 24 [0.2 to 24]
  Day 1, crossover treatment | 0 [0 to 1] | 0 [0 to 24]
  Day 7, crossover treatment | 0 [0 to 1] | 1 [0 to 24]
  Month 1, crossover treatment | 0.1 [0 to 24] | 3 [0 to 24]
  Month 2, crossover treatment | 1 [0 to 24] | 1 [0 to 24]
  Month 3, crossover treatment | 0 [0 to 24] | 10 [0 to 24]
  Month 4, crossover treatment | 0.2 [0 to 24] | 24 [0.1 to 24]
  Month 12, initial | 1 [0 to 24] | 1 [0 to 24]

11. Secondary Outcome: Non-painful Phantom Sensations Frequency
Description: Sensations that feel to emanate from the missing limb, but are not described as pain. The frequency is the number of times this is experienced in the previous 72 hours.
  To read the results: for the group that received cryoneurolysis initially followed by sham for the crossover treatment, "initial" Days 1 - Month 4 provide the results for those receiving cryoneurolysis while "crossover" Days 1 - Month 4 provide the results for those receiving sham treatment. This is reversed for the other treatment group that received sham initially followed by cryoneurolysis for the crossover treatment.
Time Frame: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Occurrences
Groups:
- Cryoneurolysis Initially; Sham Crossover Treatment: Initial treatment: Cryoneurolysis of the femoral and sciatic nerves (or their distal counterparts) in the residual limb: The cryoneurolysis device will be triggered using 3 cycles of 2-minute gas activation separated by 1-minute defrost periods. For active probes, the nitrous oxide will be deployed to the tip where a drop in temperature to -70°C will result in cryoneurolysis.
  Crossover treatment: Sham cryoneurolysis of the femoral and sciatic nerves (or their distal counterparts) in the residual limb: The cryoneurolysis device will be triggered using 3 cycles of 2-minute gas activation separated by 1-minute defrost periods. However, for sham probes, the nitrous oxide is not deployed to the tip and therefore there is no drop in temperature resulting in cryoneurolysis.
- Sham Comparator Initially; Cryoneurolysis Crossover Treatment: Initial treatment: Sham cryoneurolysis of the femoral and sciatic nerves (or their distal counterparts) in the residual limb: The cryoneurolysis device will be triggered using 3 cycles of 2-minute gas activation separated by 1-minute defrost periods. However, for sham probes, the nitrous oxide is not deployed to the tip and therefore there is no drop in temperature resulting in cryoneurolysis.
  Crossover treatment: Cryoneurolysis of the femoral and sciatic nerves (or their distal counterparts) in the residual limb: The cryoneurolysis device will be triggered using 3 cycles of 2-minute gas activation separated by 1-minute defrost periods. For active probes, the nitrous oxide will be deployed to the tip where a drop in temperature to -70°C will result in cryoneurolysis.
Arm/Group | Cryoneurolysis Initially; Sham Crossover Treatment | Sham Comparator Initially; Cryoneurolysis Crossover Treatment
Number analyzed (Participants) | 71 | 73
Occurrences
  Baseline (Day 0) | 24 [5 to 24] | 24 [4 to 24]
  Day 1, initial treatment | 0 [0 to 24] | 1 [0 to 24]
  Day 7, initial treatment | 9 [0 to 24] | 24 [0 to 24]
  Month 1, initial treatment | 12 [0 to 24] | 24 [0 to 24]
  Month 2, initial treatment | 10 [0 to 24] | 24 [0 to 24]
  Month 3, initial treatment | 24 [0 to 24] | 24 [0 to 24]
  Month 4, initial treatment | 24 [0 to 24] | 24 [0 to 24]
  Day 0, crossover treatment | 24 [2 to 24] | 24 [5 to 24]
  Day 1, crossover treatment | 0 [0 to 24] | 0 [0 to 24]
  Day 7, crossover treatment | 0 [0 to 24] | 0 [0 to 24]
  Month 1, crossover treatment | 2 [0 to 24] | 24 [0 to 24]
  Month 2, crossover treatment | 14 [0 to 24] | 0 [0 to 24]
  Month 3, crossover treatment | 2 [0 to 24] | 24 [0 to 24]
  Month 4, crossover treatment | 3 [0 to 24] | 24 [0 to 24]
  Month 12, initial | 0 [0 to 24] | 0 [0 to 24]

12. Secondary Outcome: Non-painful Phantom Sensations Duration
Description: Sensations that feel to emanate from the missing limb, but are not described as pain. The duration is the average duration of each experience over the previous 72 hours.
  To read the results: for the group that received cryoneurolysis initially followed by sham for the crossover treatment, "initial" Days 1 - Month 4 provide the results for those receiving cryoneurolysis while "crossover" Days 1 - Month 4 provide the results for those receiving sham treatment. This is reversed for the other treatment group that received sham initially followed by cryoneurolysis for the crossover treatment.
Time Frame: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Cryoneurolysis Initial Treatment; Sham Crossover Treatment | Sham, Then Optional Crossover Cryoneurolysis
Number analyzed (Participants) | 71 | 73
hours
  Baseline (Day 0) | 24 [1 to 24] | 24 [0 to 24]
  Day 1, initial treatment | 0 [0 to 24] | 0 [0 to 24]
  Day 7, initial treatment | 1 [0 to 24] | 24 [0 to 24]
  Month 1, initial treatment | 2 [0 to 24] | 24 [0 to 24]
  Month 2, initial treatment | 2 [0 to 24] | 24 [0 to 24]
  Month 3, initial treatment | 24 [0 to 24] | 24 [0 to 24]
  Month 4, initial treatment | 24 [0 to 24] | 24 [0 to 24]
  Day 0, crossover treatment | 24 [0 to 24] | 24 [0 to 24]
  Day 1, crossover treatment | 0 [0 to 24] | 0 [0 to 24]
  Day 7, crossover treatment | 0 [0 to 24] | 0 [0 to 24]
  0Month 1, crossover treatment | 0 [0 to 24] | 0 [0 to 24]
  Month 2, crossover treatment | 12.5 [0 to 24] | 0 [0 to 24]
  Month 3, crossover treatment | 2 [0 to 24] | 24 [0 to 24]
  Month 4, crossover treatment | 2 [0 to 24] | 24 [0 to 24]
  Month 12, initial | 0 [0 to 24] | 0 [0 to 24]

13. Secondary Outcome: Residual Limb Pain Frequency
Description: Pain that originates from a part of the injured limb that remains intact. The frequency is the number of times residual pain is experienced in the previous 72 hours.
  To read the results: for the group that received cryoneurolysis initially followed by sham for the crossover treatment, "initial" Days 1 - Month 4 provide the results for those receiving cryoneurolysis while "crossover" Days 1 - Month 4 provide the results for those receiving sham treatment. This is reversed for the other treatment group that received sham initially followed by cryoneurolysis for the crossover treatment.
Time Frame: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Occurrences
Arm/Group | Cryoneurolysis Initial Treatment; Sham Crossover Treatment | Sham Comparator Initially; Cryoneurolysis Crossover Treatment
Number analyzed (Participants) | 71 | 73
Occurrences
  Baseline (Day 0) | 5 [0 to 24] | 12 [0 to 24]
  Day 1, initial treatment | 0 [0 to 20] | 0 [0 to 6]
  Day 7, initial treatment | 0 [0 to 24] | 0 [0 to 24]
  Month 1, initial treatment | 0 [0 to 24] | 0 [0 to 24]
  Month 2, initial treatment | 0 [0 to 24] | 0 [0 to 24]
  Month 3, initial treatment | 0 [0 to 24] | 0 [0 to 24]
  Month 4, initial treatment | 2 [0 to 24] | 3 [0 to 24]
  Day 0, crossover treatment | 3.5 [1 to 24] | 6 [0 to 24]
  Day 1, crossover treatment | 0 [0 to 3] | 0 [0 to 0.5]
  Day 7, crossover treatment | 0 [0 to 24] | 0 [0 to 24]
  Month 1, crossover treatment | 1 [0 to 24] | 3 [0 to 24]
  Month 2, crossover treatment | 0 [0 to 24] | 3 [0 to 24]
  Month 3, crossover treatment | 0 [0 to 2] | 0 [0 to 24]
  Month 4, crossover treatment | 0 [0 to 21] | 1 [0 to 24]
  Month 12, initial | 0 [0 to 6] | 0 [0 to 24]

14. Secondary Outcome: Residual Limb Pain Duration
Description: Pain that originates from a part of the injured limb that remains intact. The duration is the average number of hours that residual pain was experienced each episode in the previous 72 hours.
  To read the results: for the group that received cryoneurolysis initially followed by sham for the crossover treatment, "initial" Days 1 - Month 4 provide the results for those receiving cryoneurolysis while "crossover" Days 1 - Month 4 provide the results for those receiving sham treatment. This is reversed for the other treatment group that received sham initially followed by cryoneurolysis for the crossover treatment.
Time Frame: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Cryoneurolysis Initial Treatment; Sham Crossover Treatment | Sham Comparator Initially; Cryoneurolysis Crossover Treatment
Number analyzed (Participants) | 71 | 73
hours
  Baseline (Day 0) | 24 [2 to 24] | 24 [1 to 24]
  Day 1, initial treatment | 1 [0 to 24] | 15 [0 to 24]
  Day 7, initial treatment | 1 [0 to 24] | 15 [0 to 24]
  Month 1, initial treatment | 2 [0 to 24] | 1 [0 to 24]
  Month 2, initial treatment | 12 [0 to 24] | 24 [0 to 24]
  Month 3, initial treatment | 1 [0 to 24] | 24 [0 to 24]
  Month 4, initial treatment | 24 [0 to 24] | 24 [1 to 24]
  Day 0, crossover treatment | 3 [0 to 24] | 4.5 [0.5 to 24]
  Day 1, crossover treatment | 0 [0 to 24] | 0.5 [0 to 24]
  Day 7, crossover treatment | 0 [0 to 24] | 24 [0 to 24]
  Month 1, crossover treatment | 0.3 [0 to 24] | 24 [0 to 24]
  Month 2, crossover treatment | 0.1 [0 to 24] | 24 [1 to 24]
  Month 3, crossover treatment | 0 [0 to 24] | 24 [0 to 24]
  Month 4, crossover treatment | 0.8 [0 to 24] | 24 [1 to 24]
  Month 12, initial | 1 [0 to 24] | 24 [1 to 24]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Cryoneurolysis | Sham Comparator
All-Cause Mortality (participants affected / at risk) | 1/120 | 1/115
Serious Adverse Events (participants affected / at risk) | 1/120 | 1/115
Other Adverse Events (participants affected / at risk) | 0/120 | 0/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cryoneurolysis (N=120) | Sham Comparator (N=115)
Dementia of unknown origin (Nervous system disorders) | 0 (0) | 1 (1) — One participant developed dementia of unknown etiology within the 6 months following his initial treatment per an adult child's report.
fall (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Three months following the active crossover treatment the participant fell while climbing stairs and fractured a clavicle which required three subsequent surgical fixation procedures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-05): https://cdn.clinicaltrials.gov/large-docs/67/NCT03449667/Prot_SAP_000.pdf